CLINICAL TRIAL: NCT02912793
Title: A Phase I/II Study to Evaluate the Safety and PK of iv Trappsol Cyclo (HP-β-CD) in Patients With Niemann-Pick Disease Type C NPC-1 and the Pharmacodynamic Effects of Treatment Upon Markers of Cholesterol Metabolism and Clinical Outcomes
Brief Title: Safety and Efficacy of Intravenous Trappsol Cyclo (HPBCD) in Niemann-Pick Type C Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cyclo Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CTD-TCNP-201
Record Dates: First submitted 2016-08-19; First posted 2016-09-23 (Estimated); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: Niemann-Pick Disease, Type C1
MeSH Terms: conditions — Niemann-Pick Disease, Type C | interventions — 2-Hydroxypropyl-beta-cyclodextrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hydroxypropyl-beta-cyclodextrin IV 1500 mg/kg (Active Comparator): Hydroxypropyl-beta-cyclodextrin administered by slow IV infusion for 8h every 2 weeks
  Interventions: Drug: Hydroxypropyl-beta-cyclodextrin
- Hydroxy-propyl-beta-cyclodextrin IV 2000 mg/kg (Active Comparator): Hydroxypropyl-beta-cyclodextrin administered by slow IV infusion for 8h every 2 weeks
  Interventions: Drug: Hydroxypropyl-beta-cyclodextrin
- Hydroxypropyl-beta-cyclodextrin IV 2500 mg/kg (Active Comparator): Hydroxypropyl-beta-cyclodextrin administered by slow IV infusion for 8h every 2 weeks
  Interventions: Drug: Hydroxypropyl-beta-cyclodextrin

INTERVENTIONS:
Drug: Hydroxypropyl-beta-cyclodextrin — Used in the treatment of Niemann-Pick C1
  Other Names: Trappsol Cyclo

SUMMARY:
This research study is being conducted to find out whether Trappsol® Cyclo™, an experimental treatment for people with Niemann-Pick disease Type C1 (NPC-1) is safe at 3 different dose levels and what effects it has on people who have this condition. NPC-1 is caused by a defect in a protein which is important for the transport of fatty substances like cholesterol out of cells. Without this protein, fats build up in the cells ultimately leading to organ damage. The way in which this experimental treatment works is not fully understood but laboratory experiments have shown that it can potentially remove cholesterol build up from the cells in people who have NPC-1. Approximately 12 patients will be asked to take part in this research study for up to 56 weeks in total. recruitment is expected to take 9 months.Patients who take part will receive treatment by an intravenous infusion every two weeks. The study will look at what the body does to the drug as well as what the drug does to the body by taking and examining blood and urine samples. Samples of Cerebrospinal fluid (CSF) are also taken by lumbar puncture during and following the first treatment dose. Patients will also have their hearing tested, be asked questions by their doctor as well completing questionnaires to help assess any changes in their condition during treatment. Optional assessments patients can choose to take part in include liver biopsies, additional lumbar punctures for CSF.examinations to see if the drug is affecting these. This study is being sponsored and funded by CTD holdings INC. It is planned to be run in the UK, Italy, and Sweden.

DETAILED DESCRIPTION:
The planned study has been designed as a Phase I/II, double-blind, randomised, multi-centre, parallel group study based on information and data available from the administration of Trappsol Cyclo via compassionate/named patient use in patients with NPC-1, and data on other cyclodextrin products in the scientific literature.

The study is comprised of two stages. The primary objective of Stage 1 is to compare the plasma pharmacokinetics of three different doses of IV Trappsol Cyclo in the prevention /delay of NPC-1 progression.Secondary objectives include investigation of the Hydroxypropyl Beta Cyclodextrin (HP-β-CD) effect of three different doses of IV Trappsol Cyclo upon serum and lymphocytic markers of cholesterol metabolism (Stages 1 and 2) and evaluation of concentrations in the cerebrospinal fluid (CSF) following intravenous (IV) administration (Stage 1), evaluation of the impact of treatment upon measures of neurological function including ataxia, aphasia and saccadic eye movements, and the impact of treatment upon behavioural aspects of NPC-1 (Stage 2).

It is planned to recruit a total of 12 patients to the study. Patients will be randomised 1:1:1 to one of the three dose levels (1500 mg/kg, 2000 mg/kg or 2500 mg/kg; four patients per dose level). Treatment will be administered every two weeks by slow IV infusion at a concentration of 250 mg/mL over 8 hours. Patients completing Stage 1 of the study will continue into Stage 2 and receive treatment for 48 weeks. Patients who withdraw prior to completion of the initial pharmacokinetic (PK) and pharmacodynamics (PD) assessments will be replaced.

The design of the proposed study thus enables early assessment of biochemical markers of response but allows for a sufficient dosing duration to enable the effectiveness of Trappsol in NPC-1 to be assessed.

As miglustat is an approved treatment for NPC-1 in the EU, with an established efficacy and safety profile, it would be unethical to exclude patients receiving miglustat therapy from the study, given that the study itself will also be conducted at sites in Europe. However, it is planned to balance randomisation across the treatment groups for its use.

The maximum dose proposed for this study is below the maximum dose for which long term clinical data is available in 2 patients (2800 mg/kg weekly for 3-5 years). Although individual clinicians have not always utilised an escalating rate of infusion, the reports of infusion related reactions in three patients suggest that this is an appropriate clinical strategy to mitigate the risk of such events and is consistent with dosing administration for other therapeutic agents. In the proposed study, treatment will be administered less frequently than has been undertaken in compassionate use. This longer dosing interval is supported by nonclinical data comparing the metabolism of cholesterol in non-human species with that in man; although a once weekly dosing interval was initially studied in man based on data in the mouse, HP-β-CD cholesterol metabolism/turnover in the mouse is 13-fold higher than in man which, in NPC-1, likely translates into a 13-fold slower accumulation of cholesterol in human cells compared with those of the mouse.Therefore, it is theorised that, given the slower cholesterol metabolism in humans, the dosing interval could be much less frequent in man than in mouse; however, based on what is known about cholesterol metabolism in humans and the pharmacokinetic and pharmacodynamic effect of HP-β-CD in the mouse, a dosing interval of 2 weeks in man is likely to be well within the therapeutic dosing interval and also minimises the amount of infusions required to be administered.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of NPC-1 defined as one of the following

   * Two NPC-1 mutations on genotyping
   * One NPC-1 mutation and positive filipin staining (current or prior)
   * Vertical supranuclear gaze palsy [VSNGP] plus either ≥ one NPC-1 mutation or positive filipin staining and no NPC-2 mutations
2. NIH NPC Severity Score <30 and with no more than 4 individual domains with a score ≥ 3.
3. Age range: 2 years upwards

   * Inclusion of the first three paediatric patients will be restricted to individuals aged ≥ 5 years. Once the first three paediatric patients have safely completed stage 1, study entry will be open to all ages ≥2 years as per the protocol
4. Negative pregnancy test for females of child bearing potential
5. Written, informed consent

   -

Exclusion Criteria:

1. The presence of NPC-2 mutations on genotyping
2. Previous receipt of cyclodextrin therapy
3. Lanksy score < 50 if aged ≤16 or Karnofsky score < 40 if aged > 16.
4. Inability to comply with the proposed protocol assessments
5. Concurrent treatment with any type of cholesterol lowering agents such as statins, fibrates, ezetimibe
6. Concurrent medical conditions representing a contraindication to any of the study medications
7. Stage 3 renal impairment or worse as indicated by eGFR< 60mL/min using the MDRD equation
8. Clinical evidence of acute liver disease including symptoms of jaundice or right upper quadrant pain or INR >1. 8
9. Involvement in another interventional clinical trial within the previous 6 months
10. Weight >100 kg
11. Females of childbearing potential who are not willing to use a method of highly effective contraception (hormonal contraception, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomised partner, or true abstinence) during the study and the follow-up period. True abstinence can only be in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), declaration of abstinence for the duration of a trial, and withdrawal are not acceptable methods of contraception.
12. Females who are breastfeeding

    -

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-03-03 (Actual)

PRIMARY OUTCOMES:
To evaluate the plasma the Maximum Concentration (C max) of 3 doses of Trappsol by measurement of plasma levels | 0,2,4,6,& 8 hours (h) after the start of the IV infusion of Trappsol and 0.5,1,2,4,8 & 12 h after the end of the infusion
  To evaluate plasma PK of Trappsol by comparison of Maximum Concentration (Cmax ) of the three doses
To evaluate the Time to Maximum Concentration ( Tmax) of 3 doses of Trappsol by measurement of plasma levels | 0,2,4,6,& 8h after the start of IV infusion of Trappsol and 0.5,1,2,4,6 &12h after the end of infusion
  To evaluate the plasma PK of Trappsol by comparison of the Tmax of three doses
To evaluate the Volume of Distribution of Trappsol by measurement of plasma levels | ),2,4,6 & 8 h after the start of the IV infusion of Trappsol and 0.5,1,2,4,8,&12 h after the end of the infusion
  To evaluate the plasma PK of Trappsol by comparison of the Volume of Distribution of three doses
To evaluate the elimination half-life of Trappsol by measurement of plasma levels | 0,2,3,6 & 8h after the start of IV infusion of Trappsol and 0.5,1,2,4,8 &12h after the end of infusion
  To evaluate the PK of Trappsol by comparison of the Elimination half-lives of three doses

SECONDARY OUTCOMES:
Markers of cholesterol metabolism | Screening,Days1,2,3,5,8,Weeks 2,4,8,10,12,14,16,18,20,24,28,32,36,40,44,48 and follow-up
  To investigate the effect of 3 different doses of intravenous Trappsol in patients upon serum and lymphocytic markers of cholesterol metabolism in patients with NPC-1
CSF levels of HP-β-CD | Pre then 4,8,and 12h after the start of the initial infusion
  To evaluate HP-β-CD concentrations in CSF following intravenous administration of Trappsol in patients with NPC-1 to determine if the drug crosses the blood brain barrier
Number of patients with treatment-related adverse events as assessed by CTCAE ( version 4.03) | Screening,Days1,2,3,4,6,8,Week 2,4,6,8,10,12,14,16,18,20,22,24,26,28,30,32,34,36,38,40,42,44,46,48 and follow-up
  Events will be gathered by spontaneous reporting, clinical observation and laboratory tests including standard audiology tests and auditory evoked potential to assess hearing
Abdominal ultrasound | Baseline 12,24,36 and 48 weeks
  Change from baseline in hepatic and splenic morphology
The proportion of patients with a reduction from baseline in the NIH NPC severity scale | Baseline and 48weeks
  Reduction of one point in two or more domains
Top evaluate the impact of treatment on ataxia | Screening, baseline and weeks 12,18,36 and 48
  Ataxia will be rated using the Scale for the assessment and rating of ataxia (SARA) in patients where age and cognitive function allow it.
To evaluate the effect of treatment on fine motor skills | Screening, baseline and weeks 12,18,36 and 48
  Motor skills will be assessed by the bead-threading test in patients where age and cognitive function allow it
To evaluate the effect of treatment on saccadic eye movements | Screening, baseline and weeks 12,18,36 and 48
  Changes in saccadic eye movements will be assessed by clinical observation.
To evaluate cognitive impairment | Screening, baseline and weeks 12,18,36 and 48
  Changes in cognitive impairment will be assessed using the Mini Mental Scale ( MMS) in patients where age and cognitive function allow it.

OTHER OUTCOMES:
Change from baseline in hepatic fractionated cholesterol | Baseline , day 2 and 48weeks
  To investigate the impact of treatment on cholesterol handling by the liver
Exploratory measures of potential CSF Biomarkers | Baseline, weeks 24and 48
  To investigate the impact of treatment upon CSF markers of NPC-1 disease

CONTACTS AND LOCATIONS:
Overall Officials: Reena Sharma, MB BS, Principal Investigator — Salford Royal Foundation NHS Trust,
Locations (5):
- Israel (2):
  - Soroka Mc, Beersheba, Rager Blvd
  - HaeMek MC, Afula
- Karolinska Trial Alliance, Solna, Huddinge, Sweden
- United Kingdom (2):
  - Salford Royal Hospital, Salford, Greater Manchester
  - Leonard Wolfson Experimental Neurology Centre, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Battisti C, Tarugi P, Dotti MT, De Stefano N, Vattimo A, Chierichetti F, Calandra S, Federico A. Adult onset Niemann-Pick type C disease: A clinical, neuroimaging and molecular genetic study. Mov Disord. 2003 Nov;18(11):1405-9. doi: 10.1002/mds.10541. PMID 14639697
- [Background] Coussement W, Van Cauteren H, Vandenberghe J, et al. Toxicological profile of Hydroxypropyl-beta-cyclodextrin (HPBCD) in laboratory animals. In: Minutes of the Fifth International Symposium on cyclodextrins; 28-30 March 1990; Paris, France: Editions de Santé; 1990 p. 522-4.
- [Background] Fischer D, Stewart AL, Bloch DA, Lorig K, Laurent D, Holman H. Capturing the patient's view of change as a clinical outcome measure. JAMA. 1999 Sep 22-29;282(12):1157-62. doi: 10.1001/jama.282.12.1157. PMID 10501119
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Giese AK, Mascher H, Grittner U, Eichler S, Kramp G, Lukas J, te Vruchte D, Al Eisa N, Cortina-Borja M, Porter FD, Platt FM, Rolfs A. A novel, highly sensitive and specific biomarker for Niemann-Pick type C1 disease. Orphanet J Rare Dis. 2015 Jun 17;10:78. doi: 10.1186/s13023-015-0274-1. PMID 26082315
- [Background] Gould S, Scott RC. 2-Hydroxypropyl-beta-cyclodextrin (HP-beta-CD): a toxicology review. Food Chem Toxicol. 2005 Oct;43(10):1451-9. doi: 10.1016/j.fct.2005.03.007. Epub 2005 Apr 19. PMID 16018907
- [Background] Greer WL, Dobson MJ, Girouard GS, Byers DM, Riddell DC, Neumann PE. Mutations in NPC1 highlight a conserved NPC1-specific cysteine-rich domain. Am J Hum Genet. 1999 Nov;65(5):1252-60. doi: 10.1086/302620. PMID 10521290
- [Background] Kamper SJ, Maher CG, Mackay G. Global rating of change scales: a review of strengths and weaknesses and considerations for design. J Man Manip Ther. 2009;17(3):163-70. doi: 10.1179/jmt.2009.17.3.163. PMID 20046623
- [Background] King KA, Gordon-Salant S, Yanjanin N, Zalewski C, Houser A, Porter FD, Brewer CC. Auditory phenotype of Niemann-Pick disease, type C1. Ear Hear. 2014 Jan-Feb;35(1):110-7. doi: 10.1097/AUD.0b013e3182a362b8. PMID 24225652
- [Background] Liu B, Li H, Repa JJ, Turley SD, Dietschy JM. Genetic variations and treatments that affect the lifespan of the NPC1 mouse. J Lipid Res. 2008 Mar;49(3):663-9. doi: 10.1194/jlr.M700525-JLR200. Epub 2007 Dec 12. PMID 18077828
- [Background] Liu B, Turley SD, Burns DK, Miller AM, Repa JJ, Dietschy JM. Reversal of defective lysosomal transport in NPC disease ameliorates liver dysfunction and neurodegeneration in the npc1-/- mouse. Proc Natl Acad Sci U S A. 2009 Feb 17;106(7):2377-82. doi: 10.1073/pnas.0810895106. Epub 2009 Jan 26. PMID 19171898
- [Background] Mattsson N, Zetterberg H, Bianconi S, Yanjanin NM, Fu R, Mansson JE, Porter FD, Blennow K. Miglustat treatment may reduce cerebrospinal fluid levels of the axonal degeneration marker tau in niemann-pick type C. JIMD Rep. 2012;3:45-52. doi: 10.1007/8904_2011_47. Epub 2011 Sep 28. PMID 23430872
- [Background] Naureckiene S, Sleat DE, Lackland H, Fensom A, Vanier MT, Wattiaux R, Jadot M, Lobel P. Identification of HE1 as the second gene of Niemann-Pick C disease. Science. 2000 Dec 22;290(5500):2298-301. doi: 10.1126/science.290.5500.2298. PMID 11125141
- [Background] Neufeld EB, Cooney AM, Pitha J, Dawidowicz EA, Dwyer NK, Pentchev PG, Blanchette-Mackie EJ. Intracellular trafficking of cholesterol monitored with a cyclodextrin. J Biol Chem. 1996 Aug 30;271(35):21604-13. doi: 10.1074/jbc.271.35.21604. PMID 8702948
- [Background] Park WD, O'Brien JF, Lundquist PA, Kraft DL, Vockley CW, Karnes PS, Patterson MC, Snow K. Identification of 58 novel mutations in Niemann-Pick disease type C: correlation with biochemical phenotype and importance of PTC1-like domains in NPC1. Hum Mutat. 2003 Oct;22(4):313-25. doi: 10.1002/humu.10255. PMID 12955717
- [Background] Patterson MC, Vecchio D, Prady H, Abel L, Wraith JE. Miglustat for treatment of Niemann-Pick C disease: a randomised controlled study. Lancet Neurol. 2007 Sep;6(9):765-72. doi: 10.1016/S1474-4422(07)70194-1. PMID 17689147
- [Background] Patterson MC, Hendriksz CJ, Walterfang M, Sedel F, Vanier MT, Wijburg F; NP-C Guidelines Working Group. Recommendations for the diagnosis and management of Niemann-Pick disease type C: an update. Mol Genet Metab. 2012 Jul;106(3):330-44. doi: 10.1016/j.ymgme.2012.03.012. Epub 2012 May 8. PMID 22572546
- [Background] Ramirez CM, Liu B, Aqul A, Taylor AM, Repa JJ, Turley SD, Dietschy JM. Quantitative role of LAL, NPC2, and NPC1 in lysosomal cholesterol processing defined by genetic and pharmacological manipulations. J Lipid Res. 2011 Apr;52(4):688-98. doi: 10.1194/jlr.M013789. Epub 2011 Feb 2. PMID 21289032
- [Background] Schicks J, Muller Vom Hagen J, Bauer P, Beck-Wodl S, Biskup S, Krageloh-Mann I, Schols L, Synofzik M. Niemann-Pick type C is frequent in adult ataxia with cognitive decline and vertical gaze palsy. Neurology. 2013 Mar 19;80(12):1169-70. doi: 10.1212/WNL.0b013e31828869f9. Epub 2013 Feb 20. No abstract available. PMID 23427322
- [Background] Schmitz-Hubsch T, du Montcel ST, Baliko L, Berciano J, Boesch S, Depondt C, Giunti P, Globas C, Infante J, Kang JS, Kremer B, Mariotti C, Melegh B, Pandolfo M, Rakowicz M, Ribai P, Rola R, Schols L, Szymanski S, van de Warrenburg BP, Durr A, Klockgether T, Fancellu R. Scale for the assessment and rating of ataxia: development of a new clinical scale. Neurology. 2006 Jun 13;66(11):1717-20. doi: 10.1212/01.wnl.0000219042.60538.92. PMID 16769946
- [Background] Sevin M, Lesca G, Baumann N, Millat G, Lyon-Caen O, Vanier MT, Sedel F. The adult form of Niemann-Pick disease type C. Brain. 2007 Jan;130(Pt 1):120-33. doi: 10.1093/brain/awl260. Epub 2006 Sep 26. PMID 17003072
- [Background] te Vruchte D, Speak AO, Wallom KL, Al Eisa N, Smith DA, Hendriksz CJ, Simmons L, Lachmann RH, Cousins A, Hartung R, Mengel E, Runz H, Beck M, Amraoui Y, Imrie J, Jacklin E, Riddick K, Yanjanin NM, Wassif CA, Rolfs A, Rimmele F, Wright N, Taylor C, Ramaswami U, Cox TM, Hastings C, Jiang X, Sidhu R, Ory DS, Arias B, Jeyakumar M, Sillence DJ, Wraith JE, Porter FD, Cortina-Borja M, Platt FM. Relative acidic compartment volume as a lysosomal storage disorder-associated biomarker. J Clin Invest. 2014 Mar;124(3):1320-8. doi: 10.1172/JCI72835. PMID 24487591
- [Background] Trendelenburg G, Vanier MT, Maza S, Millat G, Bohner G, Munz DL, Zschenderlein R. Niemann-Pick type C disease in a 68-year-old patient. J Neurol Neurosurg Psychiatry. 2006 Aug;77(8):997-8. doi: 10.1136/jnnp.2005.086785. No abstract available. PMID 16844962
- [Background] Vance JE. Dysregulation of cholesterol balance in the brain: contribution to neurodegenerative diseases. Dis Model Mech. 2012 Nov;5(6):746-55. doi: 10.1242/dmm.010124. Epub 2012 Oct 12. PMID 23065638
- [Background] Vanier MT. Niemann-Pick disease type C. Orphanet J Rare Dis. 2010 Jun 3;5:16. doi: 10.1186/1750-1172-5-16. PMID 20525256
- [Background] Vite CH, Bagel JH, Swain GP, Prociuk M, Sikora TU, Stein VM, O'Donnell P, Ruane T, Ward S, Crooks A, Li S, Mauldin E, Stellar S, De Meulder M, Kao ML, Ory DS, Davidson C, Vanier MT, Walkley SU. Intracisternal cyclodextrin prevents cerebellar dysfunction and Purkinje cell death in feline Niemann-Pick type C1 disease. Sci Transl Med. 2015 Feb 25;7(276):276ra26. doi: 10.1126/scitranslmed.3010101. PMID 25717099
- [Background] Welford RW, Garzotti M, Marques Lourenco C, Mengel E, Marquardt T, Reunert J, Amraoui Y, Kolb SA, Morand O, Groenen P. Plasma lysosphingomyelin demonstrates great potential as a diagnostic biomarker for Niemann-Pick disease type C in a retrospective study. PLoS One. 2014 Dec 5;9(12):e114669. doi: 10.1371/journal.pone.0114669. eCollection 2014. PMID 25479233
- [Background] Weyer A, Abele M, Schmitz-Hubsch T, Schoch B, Frings M, Timmann D, Klockgether T. Reliability and validity of the scale for the assessment and rating of ataxia: a study in 64 ataxia patients. Mov Disord. 2007 Aug 15;22(11):1633-7. doi: 10.1002/mds.21544. PMID 17516493
- [Background] Yamamoto T, Nanba E, Ninomiya H, Higaki K, Taniguchi M, Zhang H, Akaboshi S, Watanabe Y, Takeshima T, Inui K, Okada S, Tanaka A, Sakuragawa N, Millat G, Vanier MT, Morris JA, Pentchev PG, Ohno K. NPC1 gene mutations in Japanese patients with Niemann-Pick disease type C. Hum Genet. 1999 Jul-Aug;105(1-2):10-6. doi: 10.1007/s004399900059. PMID 10480349
- [Background] Yanjanin NM, Velez JI, Gropman A, King K, Bianconi SE, Conley SK, Brewer CC, Solomon B, Pavan WJ, Arcos-Burgos M, Patterson MC, Porter FD. Linear clinical progression, independent of age of onset, in Niemann-Pick disease, type C. Am J Med Genet B Neuropsychiatr Genet. 2010 Jan 5;153B(1):132-40. doi: 10.1002/ajmg.b.30969. PMID 19415691
- [Derived] Sharma R, Hastings C, Staretz-Chacham O, Raiman J, Paucar M, Spiegel R, Murray B, Hurst B, Liu B, Kjems L, Hrynkow S. Long-term administration of intravenous Trappsol(R) Cyclo (HP-beta-CD) results in clinical benefits and stabilization or slowing of disease progression in patients with Niemann-Pick disease type C1: Results of an international 48-week Phase I/II trial. Mol Genet Metab Rep. 2023 Jun 29;36:100988. doi: 10.1016/j.ymgmr.2023.100988. eCollection 2023 Sep. PMID 37670901